CLINICAL TRIAL: NCT04430556
Title: Study on the Brain Hippocampal Volume, Cortisol and C-reactive Protein Levels Relationship With Anxious Symptoms in Major Depressive Patients
Brief Title: Brain Hippocampal Volume Relationship With Anxious Symptoms in Major Depressive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Instituto de Información e Investigación en Salud Mental A. C. (Unknown)
Responsible Party: Principal Investigator, José Alfonso Ontiveros Sánchez De la Barquera, Associate Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PS18-00016
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder; Anxiety Disorders
Keywords: major depressive disorder; hippocampal volume; cortisol; c-reactive protein; brain metabolites; MRI; anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volumetric changes in response to sertraline or escitalopram (Other)
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Sertraline will be started in all patients, unless it is contraindicated, in this case, Escitalopram will be indicated.

SUMMARY:
The objective of this transversal study is to determine if there is a difference in the volume of the hippocampus with the degree of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* First-time patients, without prior antidepressant treatment that meet the diagnostic criteria of DSM 5 for major depressive disorder.
* Patients who meet the current major depressive disorder criteria in the MINI interview.
* Patients who signed the informed consent for the investigation.

Exclusion Criteria:

* Patients presenting insufficient data in the MINI interview for current major depression.
* Patients diagnosed with intellectual development disorder, by clinic.
* Patients with diagnosis of the schizophrenic spectrum, bipolar disorder, autism spectrum disorder, post-traumatic stress disorder and obsessive-compulsive disorder by clinic and / or by the MINI interview.
* Patients with contraindications for MRI.
* Patients with serious or unstable medical problems.
* Patients undergoing some legal procedure.
* Patients with difficulties in understanding the interview or completing the assessment instruments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Response on Hamilton Anxiety Rating Scale | Change from baseline to week 8
  The Hamilton Anxiety Rating Scale and its correlation with hippocampal size

SECONDARY OUTCOMES:
Response on Clinical Global Impression-Improvement | Change from baseline to week 8
  Difference between baseline and final score
Response on Hamilton Depression Rating Scale | Change from baseline to week 8
  Difference between baseline and final score
Response on Montgomery-Asberg Scale for Depression | Change from baseline to week 8
  Difference between baseline and final score
Response on Columbia Scale for Suicidality | Change from baseline to week 8
  Difference between baseline and final score
Response on State-Trait Depression Inventory | Change from baseline to week 8
  Difference between baseline and final score
Response on Beck Anxiety Inventory | Change from baseline to week 8
  Difference between baseline and final score
Response on EQ-5D | Change from baseline to week 8
  Difference between baseline and final score

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Ontiveros Sanchez de la Barquera, MD, PhD, Study Chair — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico